CLINICAL TRIAL: NCT00356330
Title: Study to Evaluate Safety of Cardiac Pacemakers in MR Imaging at 3T Tesla
Brief Title: Safety of Cardiac Pacemakers in 3 Tesla MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Other Study IDs: 116/06
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Heart Diseases
Keywords: pacemaker; magnetic resonance imaging; safety
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
To evaluate short-term and long-term effects by MR imaging at 3T on the technical and functional status of cardiac pacemakers.

DETAILED DESCRIPTION:
Recently, a shift could be observed from cardiac pacemakers being an absolute contraindication to being a relative contraindication for MR imaging at 1.5 Tesla, depending on a patient-per-patient risk-benefit-evaluation, which includes an urgent clinical need for MR imaging (other imaging modalities non-conclusive) and co-morbidities (especially cardiac co-morbidities). At the same time, MR imaging at 3 Tesla is evolving from a research application only to an important imaging modality today.

Using the improved signal-to-noise-ratio, high field MR-Systems with a field strength of 3 Tesla offer a variety of diagnostic advantages to 1.5 Tesla systems. These advantages lead to a higher sensitivity and specificity in diagnosing, foremost neurological, disorders.

In this study, we evaluate the safety of MR imaging of the brain in patients with cardiac pacemakers at 3T.

ELIGIBILITY:
Inclusion Criteria:

* Urgent need for an MRI examination
* Stable pacemaker physical parameters

  * Battery voltage > 2.7 V
  * Battery impedance < 2000 Ohm
  * Battery estimated remaining lifetime > 6 months
  * Lead impedances 200-2000 Ohm
* Stable pacing parameters

  * Pacing capture threshold <2.5V at a pulse duration of 0.4ms
  * Sensing > 5mV
* Minimum 3 months since pacemaker and lead implantation

Exclusion Criteria:

* History of ventricular tachycardia (VT) or ventricular fibrillation
* Unstable angina
* Myocardial infarction within the previous 3 months
* Cardiothoracic surgery within the previous 3 months
* Presence of an abdominal pacemaker with lead length > 70 cm
* Presence of MRI incompatible bioimplants or other MRI incompatible materials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Sommer, MD, Principal Investigator — University of Bonn, Department of Radiology
Locations (1):
- University of Bonn, Department of Radiology, Bonn, North Rhine-Westphalia, Germany